CLINICAL TRIAL: NCT06001827
Title: SAVE-FistulaS: the SelfWrap-Assisted ArterioVEnous Fistulas Study
Acronym: SAVE-FistulaS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VenoStent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VENO-CIP002
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases; End Stage Renal Disease; Arteriovenous Fistula; Hemodialysis Access Failure; ESRD; Vascular Access Complication; Renal Failure; Catheter Complications; Catheter Dysfunction; Renal Insufficiency
Keywords: Vascular Surgery; Vascular Access; Nephrology; Bioabsorbable; Perivascular Wrap; External Support; Hemodialysis; Dialysis; Chronic Kidney Disease; End Stage Renal Disease; Arteriovenous Fistula; AVF
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Arteriovenous Fistula; Renal Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Arm (Experimental): Treated with SelfWrap Bioabsorbable Perivascular Wrap during AVF creation surgery
  Interventions: Device: SelfWrap Bioabsorbable Perivascular Wrap
- Control Arm (Sham Comparator): AVF creation surgery without any intervention (untreated AVF control, or standard of care)
  Interventions: Procedure: Untreated AVF Control

INTERVENTIONS:
Device: SelfWrap Bioabsorbable Perivascular Wrap — SelfWrap is applied during arteriovenous fistula (AVF) creation surgery. It provides mechanical support to improve maturation and patency of AVFs.
  Other Names: SelfWrap
  Arms: Treatment Arm
Procedure: Untreated AVF Control — AVF creation surgery without any intervention
  Other Names: Standard of Care
  Arms: Control Arm

SUMMARY:
This is a prospective, randomized, multi-center clinical trial for chronic kidney disease (CKD) patients referred for creation of a new arteriovenous fistula (AVF) in order to assess the safety and effectiveness of SelfWrap, a bioabsorbable perivascular wrap.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, double-arm, single-blind, evaluator-blinded clinical trial for CKD patients referred for creation of a new arteriovenous fistula (AVF). This study will involve approximately 200 participants from up to 25 investigational sites, randomized 1:1 to treatment with the SelfWrap or the untreated AVF control (i.e. standard of care, SOC). Participants will be followed for a duration of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Referred for creation of a new AVF
* Willing and able to comply with study requirements, communicate with the study team, and attend follow up visits over a period of 36 months

Exclusion Criteria:

* Planned index procedure to revise or repair an existing fistula
* Target artery inner diameter < 2.0 mm, as measured by ultrasound while the target arm is under tourniquet pressure and anesthesia
* Target vein inner diameter < 2.0 mm, as measured by ultrasound while the target arm is under tourniquet pressure and anesthesia
* Significant (at least 50%) stenosis at the target vein on the side of surgery (between the planned anastomosis site and the axillary vein), as diagnosed by preoperative ultrasound
* Known central venous stenosis of at least 50% on the side of surgery
* Presence of a stent or a stent graft within the access circuit
* Known or suspected coagulation disorder that, in the opinion of the Investigator, puts too much risk on the patient for AVF creation
* Known or suspected active infection at the time of surgery
* Congestive heart failure NYHA class 4
* Prior steal on the side of surgery;
* Enrolled in another investigational drug, device, or biological study, or was previously enrolled in this study
* Life expectancy less than 12 months
* Expected to undergo kidney transplant surgery within 6 months of enrollment
* Expected to undergo home hemodialysis
* Females of childbearing potential (premenopausal and not surgically sterile) without documented current negative pregnancy test at screening
* Presence of a comorbid condition that, in the opinion of the Investigator, may significantly confound the collection of safety and efficacy data in this study
* Unwillingness or inability to give consent and/or comply with the study follow up schedule
* Any health condition, which in the opinion of the Investigator, would interfere with the safety of the participant or the participant's ability to comply with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Unassisted Maturation by 180 days | Assessed at up to 6 months
  A participant who is either 1) on hemodialysis on or before day 150 and the AVF has been cannulated with two needles for at least 75% of dialysis sessions within any 4 consecutive week period to achieve the prescribed dialysis by the 180 day follow up, and did not require any facilitative endovascular or surgical intervention to achieve this, or 2) is not on hemodialysis on or before day 150, but ultrasound measurements by the 180 day follow up indicate a proximal arterial flow rate of at least 500 mL/min and a vein inner diameter of at least 5.0 mm at 5 - 8 cm from the anastomosis, and did not require any facilitative endovascular or surgical intervention through the 180 day follow up.
Freedom from access-related adverse events through 30 days | Assessed through 30 days
  Freedom from access-related adverse events through 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Boire, PhD, Study Director — VenoStent, Inc.
Locations (22):
- United States (22):
  - AKDHC Bullhead City, Bullhead City, Arizona
  - AKDHC Marana Surgery Center, Marana, Arizona
  - Arizona Kidney Disease & Hypertension Centers (AKDHC) Phoenix Surgery Center, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Tallahassee Research Institute, Tallahassee, Florida
  - Lutheran Medical Group, Fort Wayne, Indiana
  - Surgical Associates of Lexington, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health, Lake Success, New York
  - Surgical Specialists of Charlotte, P.A., Charlotte, North Carolina
  - WakeMed, Raleigh, North Carolina
  - MUSC Charleston, Charleston, South Carolina
  - MUSC Black River, Florence, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Medical University of South Carolina (MUSC) Orangeburg / Dialysis Access Institute, Orangeburg, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Saint David's HealthCare Partnership, L.P., LLP, Austin, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Houston Methodist Research Institute (Sugar Land), Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SAVE-FistulaS website — https://www.savefistulas.org
- See also: VenoStent website — https://www.venostent.com